CLINICAL TRIAL: NCT00966160
Title: Phase 3, Single Center, Controlled, Investigator-blinded, Randomized Matched Pair Design Study of CD4 Cell Recovery in HIV-1 Patients With Sustained Virologic Response Comparing Protease Inhibitor and Non-nucleoside Reverse Transcriptase Inhibitor Based Treatment Regimes
Brief Title: CD4 Cell Recovery in HIV-1 Patients Comparing 2 Treatment Regimes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Responsible Party: Dirk Taubert, University of Cologne
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HIV-1999-LRE
Record Dates: First submitted 2009-08-25; First posted 2009-08-26 (Estimated); Last update posted 2009-09-29 (Estimated); Status verified 2009-08

CONDITIONS: Acquired Immunodeficiency Syndrome; HIV Infections
Keywords: treatment naive
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; HIV Infections | interventions — Lopinavir; Ritonavir; lamivudine, zidovudine drug combination; efavirenz; Lamivudine; Zidovudine

STUDY DESIGN:
Who Masked: Investigator

ARMS (2):
- PI (Active Comparator): 400 mg lopinavir and 100 mg ritonavir (Kaletra capsules, Abbott Laboratories) twice daily plus 150 mg lamivudine (Epivir tablets, GlaxoSmithKline) and 300 mg zidovudine (Retrovir tablets, GlaxoSmithKline) twice daily over a 56-week run-in and a 420-week follow-up
  Interventions: Drug: Lopinavir/Ritonavir plus Lamivudine/Zidovudine
- NNRTI (Active Comparator): 600 mg efavirenz (Sustiva tablets, Bristol-Myers Squibb) once daily plus 150 mg lamivudine (Epivir tablets, GlaxoSmithKline) and 300 mg zidovudine (Retrovir tablets, GlaxoSmithKline) twice daily over a 56-week run-in and a 420-week follow-up
  Interventions: Drug: Efavirenz plus Lamivudine/Zidovudine

INTERVENTIONS:
Drug: Lopinavir/Ritonavir plus Lamivudine/Zidovudine — 400 mg lopinavir and 100 mg ritonavir (Kaletra capsules, Abbott Laboratories) twice daily plus 150 mg lamivudine (Epivir tablets, GlaxoSmithKline) and 300 mg zidovudine (Retrovir tablets, GlaxoSmithKline) twice daily over 476 weeks
  Arms: PI
Drug: Efavirenz plus Lamivudine/Zidovudine — 600 mg efavirenz (Sustiva tablets, Bristol-Myers Squibb) once daily plus 150 mg lamivudine (Epivir tablets, GlaxoSmithKline) and 300 mg zidovudine (Retrovir tablets, GlaxoSmithKline) twice daily over 476 weeks
  Arms: NNRTI

SUMMARY:
Therapy guidelines recommend the use of either the non-nucleoside reverse transcriptase inhibitor (NNRTI) efavirenz or a ritonavir-boostered protease inhibitor (PI) plus 2 nucleoside reverse transcriptase inhibitors (NRTI) as first-line treatment regimes of HIV-1 infection. Recent clinical studies suggest potential advantages of NNRTI- over PI-based regimes in therapy initiation due to lower rates of virologic failure and less metabolic side-effects. In contrast, PI regimes were claimed to cause greater increases in CD4 cell count than NNRTI regimes, which has been attributed to intrinsic antiapoptotic effects of the PI. However, it is still unclear whether the immunological response to a PI-containing regime is greater than to an NNRTI-containing regime, whether there is a difference in the extent of reduction of apoptosis between PI and NNRTI regimes and whether a difference in apoptosis is associated with a difference in CD4 cell recovery.

We conducted a controlled, long-term, random matched pair design study in HIV-1 infected individuals under sustained virologic suppression to evaluate in head-to-head comparison the clinical effects of a constant PI-based or NNRTI-based regime on CD4 cell recovery and the underlying molecular, biochemical and functional mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Recent, non-acute HIV-1 infection
* Caucasians
* BMI between 17.5 and 30 kg/m2
* CD4 count <200 cells/µl
* Plasma viral load >100,000 HIV-1 RNA copies/ml

Exclusion Criteria:

* Actual or previous antiretroviral therapy
* Acute illness
* Coinfection with HBV or HCV
* Opportunistic infection (Pneumocystis jiroveci pneumonia, Toxoplasma gondii encephalitis, Mycobacterium ssp. infection, syphilis, cryptosporidiosis, cryptococcosis, aspergillosis, cytomegalovirus infection or progressive multifocal leukoencephalopathy)
* Hepatic or renal disorder
* Severe cardiovascular disease
* Hematologic disorder
* Autoimmune disorder
* Diabetes mellitus or other severe endocrine disorder
* Malignancy
* Neurocognitive disorder
* Psychiatric disorder
* Drug or alcohol addiction
* Chronic drug use (except of blood pressure-lowering or lipid-lowering drugs or proton-pump inhibitors)
* Any acute medication within 7 days or vaccination within 30 days prior to entry
* Pregnancy or lactation

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 215 (Actual)
Dates: Start 1999-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Difference in changes of CD4 cell count between PI and NNRTI groups | 420 weeks

SECONDARY OUTCOMES:
Evolution of CD4 cell counts | 420 weeks
Molecular, biochemical and functional markers of CD4 cell apoptosis | 420 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Taubert, MD PhD, Study Director — Department of Pharmacology, University of Cologne, Germany
Locations (1):
- Medical Clinic I and Department of Pharmacology, University of Cologne, Cologne, Germany

REFERENCES:
- [Background] Riddler SA, Haubrich R, DiRienzo AG, Peeples L, Powderly WG, Klingman KL, Garren KW, George T, Rooney JF, Brizz B, Lalloo UG, Murphy RL, Swindells S, Havlir D, Mellors JW; AIDS Clinical Trials Group Study A5142 Team. Class-sparing regimens for initial treatment of HIV-1 infection. N Engl J Med. 2008 May 15;358(20):2095-106. doi: 10.1056/NEJMoa074609. PMID 18480202
- [Background] Staszewski S, Morales-Ramirez J, Tashima KT, Rachlis A, Skiest D, Stanford J, Stryker R, Johnson P, Labriola DF, Farina D, Manion DJ, Ruiz NM. Efavirenz plus zidovudine and lamivudine, efavirenz plus indinavir, and indinavir plus zidovudine and lamivudine in the treatment of HIV-1 infection in adults. Study 006 Team. N Engl J Med. 1999 Dec 16;341(25):1865-73. doi: 10.1056/NEJM199912163412501. PMID 10601505
- [Background] Badley AD, Pilon AA, Landay A, Lynch DH. Mechanisms of HIV-associated lymphocyte apoptosis. Blood. 2000 Nov 1;96(9):2951-64. PMID 11049971